CLINICAL TRIAL: NCT07191288
Title: Assessing the Acute Effects of Virtual Reality Interventions on Stress: A Four-Arm RCT
Brief Title: Assessing the Acute Effects of Virtual Reality Interventions on Stress
Acronym: VR_Stress_25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01814
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Slow Breathing
Keywords: Virtual Reality; Stress; Breathing; Biofeedback
MeSH Terms: conditions — Hypoventilation; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR-Breathing+Mystical (Experimental): Participants engage in guided slow-paced breathing using VR that provides mystical-type visual feedback.
  Interventions: Device: VR (VR-Breathing+Mystical)
- VR-Mystical (Experimental): Participants passively view the same nature scene as in the first condition (VR-Breathing+Mystical), but without guided breathing instructions (i.e., they breathe naturally).
  Interventions: Device: VR (VR-Mystical)
- Non-VR-Breathing (Experimental): Participants follow a slow-paced breathing pattern guided by a simple visual cue (expanding/contracting circle) on a standard computer screen.
  Interventions: Device: Computer (Non-VR-Breathing)
- VR-Control (Sham Comparator): To control for the effects of experiencing VR, participants will watch a neutral documentary in a video player implemented in VR.
  Interventions: Drug: VR (VR-Control)

INTERVENTIONS:
Device: VR (VR-Breathing+Mystical) — The VR-based slow-paced breathing application is designed to provide rewarding biofeedback for a specific breathing pattern characterized by prolonged exhales. As users extend their exhales, a veil of fog gradually lifts, introducing a mystical type experience. Over time, users are rewarded with a full 360-degree panoramic view of the beautiful nature scene, accompanied by relaxing music. After approximately 5 minutes of prolonged exhales, the nature scene responds to the user's breathing by slowing down, with falling snowflakes moving more slowly, further enhancing the mystical atmosphere. This intervention was designed to be visually captivating, mystically evocative, and emotionally engaging. Duration: 10 minutes.
  Arms: VR-Breathing+Mystical
Device: VR (VR-Mystical) — Users will experience the gradual unveiling of a beautiful natural landscape as the fog lifts, and eventually, the scene slows down similar to the VR Breathing+Mystical condition. However, this application does not provide any biofeedback or breathing instructions. Users are invited to passively observe the unfolding experience, immersing themselves in the environment for 10 minutes. Relaxing music accompanies the scene. This condition relies solely on the immersive and aesthetic qualities of the virtual environment to potentially induce relaxation.
  Arms: VR-Mystical
Device: Computer (Non-VR-Breathing) — In this conventional breathing intervention, participants will be instructed to follow a slow-paced breathing pattern guided by a simple visual cue (an expanding and contracting circle) displayed on a computer screen for 10 minutes. This condition is designed to guide slow-paced breathing without incorporating any rewarding elements.
  Arms: Non-VR-Breathing
Drug: VR (VR-Control) — In the control condition, participants will watch a neutral documentary for 10 minutes in VR. This condition is used to control for the effects of the immersive VR experience. It does not include any components related to guided breathing or mystical-type content, or any form of rewarding elements.
  Arms: VR-Control

SUMMARY:
A Four-Arm RCT, testing the acute effects of a Virtual Reality (VR)- based slow-paced breathing intervention on subjective and physiological markers of stress. The investigator hypothesize that combining slow breathing with immersive, mystical-type VR elements will result in the greatest stress reduction.

ELIGIBILITY:
Inclusion Criteria:

* > 60 points on the PSQ-30 out of a maximum 120-point scale in the screening
* Healthy
* Aged between 18-35
* Fluent in German

Exclusion Criteria:

* A current diagnosis of psychiatric disorders (self-reported)
* Chronic medication use (except oral contraceptives)
* Parallel participation in another medical or psychological study
* Suicidal tendencies (PHQ-9 item 9 > 0)3
* PHQ-9 score ≥ 10
* A visual impairment not corrected by glasses or contact lenses

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Subjective stress | Assessed before and after the 10-minute interventions.
  Subjective stress measured using visual analogue scales (VAS) on a computer

SECONDARY OUTCOMES:
Mood | Assessed before and after the 10-minute interventions.
  Mood measured using visual analogue scales (VAS) on a computer.
Anxiety | Assessed before and after the 10-minute interventions.
  Anxiety measured using visual analogue scales (VAS) on a computer.
Relaxation | Assessed before and after the 10-minute interventions.
  Relaxation measured using visual analogue scales (VAS) on a computer.
Electrodermal Activity | Assessed during the 10-minute interventions.
  Physiological responses measured via Electrodermal Activity.
Respiration | Assessed during the 10-minute interventions.
  Physiological responses measured via Piezoelectric Sensor (detecting variations in abdominal movement during respiration).
Blood volume pulse | Assessed during the 10-minute interventions.
  Blood volume pulse measured via Photoplethysmography.
Heart rate (variability) | Assessed during the 10-minute interventions.
  Heart rate outcomes (e.g., HR, HRV) measured via Electrocardiogram.
Perceived mysticality | Assessed after the 10-minute interventions.
  Perceived mysticality assessed using the Mystical Experience Questionnaire-30 questionnaire.
User experience | Assessed after the 10-minute interventions.
  Average user experience measured via visual analogue scales (VAS) on a computer.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Chair — University of Basel, Research Platform Molecular and Cognitive Neuroscience
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underline results in a publication will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available after publication, study protocol (including statistical analysis plan) will be made available before start of the study.
Access Criteria: All IPD (de-identified) that underline results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Request will be reviewed by the team of the principal investigator.